CLINICAL TRIAL: NCT02405663
Title: How Can Methods of Placental Delivery Affect the Amount of Blood Loss During Cesarean Section?
Brief Title: Methods of Placental Delivery and the Amount of Blood Loss During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, ahmed abdulmoneim altraigey, lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: afhsr-1-3-2015
Record Dates: First submitted 2015-03-18; First posted 2015-04-01 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Complications; Cesarean Section
Keywords: blood loss; caesarean section; placental delivery
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- manual removal group (Experimental): Group will be assigned for manual removal of the placenta as the surgeon will introduce his hand into the uterine cavity to cleave the placenta from the decidua basalis as soon as possible after the delivery of the baby by caesarean section
  Interventions: Procedure: manual removal
- cord traction group (Experimental): Group will be assigned for controlled cord traction as the surgeon do external uterine massage and gentle traction on the exposed umbilical cord to facilitate placental delivery after the delivery of the baby by caesarean section
  Interventions: Procedure: cord traction

INTERVENTIONS:
Procedure: manual removal — one of the standard procedures for placental delivery during caesarean section the surgeon will introduce his hand into the uterine cavity to cleave the placenta from the decidua basalis as soon as possible after the delivery of the baby
  Arms: manual removal group
Procedure: cord traction — one of the standard procedures for placental delivery during caesarean section the surgeon do external uterine massage and gentle traction on the exposed umbilical cord to facilitate placental delivery
  Arms: cord traction group

SUMMARY:
To compare between the effect of controlled cord traction and manual removal of the placenta on blood loss among women undergoing caesarean sections

DETAILED DESCRIPTION:
Cesarean section (CS) is one of the most commonly performed major abdominal operations in women worldwide and its rate is increasing dramatically every year.

Some of the reported short-term morbidities include hemorrhage, postoperative fever and endometritis. The method of delivering the placenta is one procedure that may contribute to an increase or decrease in the morbidity of CS.

On an average 0.5-1 liter of blood is lost during CS, many variable techniques have been tried to reduce this blood loss. Such techniques include finger splitting versus scissor cutting of incision, in situ stitching verses exteriorization and stitching of uterus , and finally spontaneous or manual removal of the placenta.

Two common methods used to deliver the placenta at CS are cord traction and manual removal.

Manual removal of the placenta which the obstetrician introduce his hand into the uterine cavity to cleave the placenta from the decidua basalis as soon as possible after the delivery of the infant and controlled cord traction in which the obstetrician do external uterine massage and gentle traction on the exposed umbilical cord to facilitate placental delivery.

Opinions differ about the best for placental delivery technique at CS. Some trials showed a reduced risk of blood loss with controlled cord traction (3) and others showed that manual removal of placenta at CS do not increase perioperative blood loss.

Authors concluded that manual delivery of the placenta was significantly associated with greater operative blood loss and greater decrease in postoperative hemoglobin levels and postpartum maternal infectious morbidity but with shorter operative time compared with spontaneous placental separation .

In addition, it is known that the blood loss at CS delivery is difficult to estimate, and numerous different methods including serial change in hematocrit (Hct), hemoglobin (Hb) level, visual estimation and the gravimetric method are described.

A low, but significant, correlation was found between visually estimated blood loss and perioperative hemoglobin change in women delivering by CS. However, hemoglobin , hematocrit levels and visual estimation are the most commonly used technique for estimating blood loss at delivery.

ELIGIBILITY:
Inclusion Criteria:

- All informed and consented women undergoing elective or emergency CS will be legible for enrollment into the study

Exclusion Criteria:

* Multiple gestation.
* Pregnancy below 34 weeks.
* Severe maternal anemia.
* Severe pre-eclampsia
* Prolonged labor.
* Prolonged rupture of the membranes with fever.
* Placental abruption.
* Placenta previa.
* Placenta accreta.
* Clotting disorders.
* Current or previous history of a significant disease including heart disease, liver, renal disorders.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
blood loss assessment after placental delivery | 12 hours
  Determine estimated blood loss after placental delivery either by cord traction or manually during caesarean section through comparing pre and postoperative hemoglobin and haematocrit measurements

SECONDARY OUTCOMES:
Placental delivery time. | 30 minutes
  time needed to deliver the placenta calculated from time of full baby delivery to the time of full placental delivery
Duration of operation | 2 hours
  time calculated from first skin incision to the time of last stitch
Need to use ecbolics | 30 minutes
  documentation of the type, the dose of different ecbolics needed to stop any possible bleeding
Need of blood transfusion | 12 hours
  documentation of the need and the amount needed of packed red blood cells packs or any other blood products if patient general condition required
Blood loss > 1000 ml | 12 hours
  counting down the cases of estimated blood loss more than 1000ml
postoperative endometritis and puerperal pyrexia | one week
  counting down the cases of puerperal pyrexia after exclusion of all other etiologies rather than endometritis

CONTACTS AND LOCATIONS:
Overall Officials: mohammed ellaithy, Principal Investigator — Ain Shams University; haytham atia, Principal Investigator — Zagazig University; nuzhat amer, Principal Investigator — Armed Forces Hospitals, Southern Region, Saudi Arabia; ahmed altraigey, Study Director — Benha University
Locations (1):
- Postpartum ward of Armed Forces Hospital, Southern Region, Khamis Mushait, 'Asir Region, Saudi Arabia